CLINICAL TRIAL: NCT03882905
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Lipid-Altering Efficacy, Safety, and Tolerability of SCH 58235 When Added to Ongoing Therapy With an HMG-CoA Reductase Inhibitor (Statin) in Patients With Primary Hypercholesterolemia, Known Coronary Heart Disease, or Multiple Cardiovascular Risk Factors
Brief Title: A Study of SCH 58235 (Ezetimibe) When Added to Ongoing Therapy With a Statin in Participants With Primary Hypercholesterolemia, Known Coronary Heart Disease, or Multiple Cardiovascular Risk Factors (P02173)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02173; MK-0653-001 (Other: Merck); SCH 58235 P02173 (Other: Schering-Plough)
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Ezetimibe; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ezetimibe: Base Study (Experimental): 10-mg tablet, oral taken once daily concomitantly with the participant' s current statin therapy for 8 weeks.
  Interventions: Drug: Ezetimibe; Drug: Statin
- Placebo: Base Study (Placebo Comparator): Placebo for ezetimibe 10-mg tablet, oral taken once daily concomitantly with the participant' s current statin therapy for 8 weeks.
  Interventions: Drug: Placebo; Drug: Statin
- Ezetimibe: Extension (Experimental): 10-mg tablet, oral taken once daily concomitantly with simvastatin for 48 weeks.
  Interventions: Drug: Ezetimibe; Drug: Simivastatin
- Placebo: Extension (Placebo Comparator): Placebo for ezetimibe tablet, oral taken once daily concomitantly with simvastatin for 48 weeks.
  Interventions: Drug: Placebo; Drug: Simivastatin

INTERVENTIONS:
Drug: Ezetimibe — 10 mg tablet, oral, once daily
  Arms: Ezetimibe: Base Study; Ezetimibe: Extension
Drug: Placebo — one tablet, oral, once daily
  Arms: Placebo: Base Study; Placebo: Extension
Drug: Simivastatin — Once daily administration at dose to be determined
  Arms: Ezetimibe: Extension; Placebo: Extension
Drug: Statin — Statin administered orally once daily at dose determined by treatment prior to enrollment by personal physician
  Arms: Ezetimibe: Base Study; Placebo: Base Study

SUMMARY:
This is a study to evaluate the lipid-altering efficacy, safety, and tolerability of ezetimibe when added to ongoing therapy with an 3-hydroxy-3-methyl-glutaryl-coenzyme A (HMG-CoA) reductase inhibitor (statin) in participants with primary hypercholesterolemia, multiple cardiovascular risk factors, or known coronary heart disease (CHD) or CHD-equivalent disease. The statin and dose in use by the participant at screening will be maintained at the same dose for the 8-week treatment phase of the study. Following the treatment, there will be a 6-week cholesterol reversibility phase to determine the rebound effect on cholesterol after ezetimibe is discontinued, but the participant is still on their statin therapy. The primary hypothesis is that the addition of ezetimibe 10 mg/day to ongoing statin monotherapy will result in a further reduction in low-density lipoprotein-cholesterol (LDL-C) compared with placebo.

The protocol was amended to include an extension for participants who complete the base study. The extension will evaluate the safety and tolerability of concomitant treatment of simvastatin with ezetimibe10 mg/day over a 1-year period. All participants in the extension will be converted from current statin to an equivalent dose of simvastatin for 6 weeks. Participants then will be randomly assigned to receive simvastatin coadministered with either with Ezetimibe 10 mg daily or matching placebo for the reminder of study.

ELIGIBILITY:
Inclusion Criteria

* Currently taking an approved and stable (for at least 6 weeks prior to screening) daily dose of a statin and by history had taken >80% of daily doses for the preceding 6 weeks
* Have a negative pregnancy test
* Agree to practice an effective barrier method of birth control during the study if of childbearing potential
* Females receiving hormonal therapy, including hormone replacement, any estrogen antagonist/agonist, or oral contraceptives, maintain a stable dose and regimen for at least 8 weeks and be willing to continue the same regimen for the duration of the study
* Must verify previous instruction on an National Cholesterol Education Program (NCEP) Step 1 diet or similar diet and must maintain a stable diet regimen for the duration of the study
* Weight stability ( ± 2 kg) for at least 6 weeks prior to entry into the study Exclusion Criteria
* History of mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy
* Previously enrolled to any study evaluating ezetimibe
* Pregnant or lactating
* Consumes greater than 14 alcoholic drinks/week
* Taking a lipid-altering agent (other than statins) in previous 6 weeks
* Taking Oral corticosteroids, unless the corticosteroids were for replacement therapy to treat pituitary/adrenal disease and were treated with a stable regimen for at least the previous 6 weeks
* Treatment with psyllium, other fiber-based laxatives, and other over-the-counter (OTC) therapies that affect serum lipids, unless treated with a stable regimen for at least 6 weeks
* Taking orlistat
* Taking cyclosporine
* Use of any investigational drugs within 30 days
* Treatment with agents with known interactions with statins including antifungal azoles (itraconazole and ketoconazole), macrolide antibiotics (erythromycin and clarithromycin) and nefazodone or with other potent agents that could significantly interfere with cytochrome P-450 system
* Congestive heart failure New York Heart Association (NYHA) Class III or IV
* Uncontrolled cardiac arrhythmias
* Myocardial infarction, coronary artery bypass surgery or angioplasty within 3 months
* Unstable or severe peripheral artery disease within 3 months
* Unstable angina pectoris
* Disorders of the hematologic, digestive or central nervous systems including cerebrovascular disease and degenerative disease that would limit study evaluation or participation
* Poorly controlled or newly diagnosed (within 3 months) diabetes mellitus, or change in antidiabetic pharmacotherapy (i.e., change in dosage [with the exception of ± 10 units of insulin] or addition of new medication) within 3 months
* Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins (i.e., secondary causes of hyperlipidemia). Clinically euthyroid participants on replacement doses of thyroid hormone are eligible for enrollment if thyroid stimulating hormone (TSH) is within the normal range
* Impaired renal function, nephrotic syndrome, or other renal disease
* Active or chronic hepatobiliary or hepatic disease
* Positive for human immunodeficiency virus (HIV)
* Cancer within the past 5 years (except for basal cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 769 (Actual)
Dates: Start 2001-01-31 (Actual); Primary Completion 2001-07-27 (Actual); Study Completion 2001-07-27 (Actual)

PRIMARY OUTCOMES:
Percentage Change from Baseline in LDL-C: Base Study | Baseline and Week 8 of Base Study
Percentage Participants with Consecutive Elevations ≥3 x Upper Limit of Normal (ULN) in Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT): Extension | up to 48 weeks (Extension)

SECONDARY OUTCOMES:
Percentage of Participants Achieving LDL-C National Cholesterol Education Program (NCEP) Adult Treatment Program II (ATP II) Target Levels: Base Study | Week 8 of Base Study
Percentage Change from Baseline in Total Cholesterol (TC) : Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in Triglycerides (TG): Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in High-density Lipoprotein-cholesterol (HDL-C) : Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in Non-HDL-C: Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in Apolipoprotein B (apoB) : Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in Apolipoprotein A-I (Apo A-I) : Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in Apolipoprotein A-II (Apo A-II) : Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in LDL-C:HDL-C Ratio: Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in Total-C:HDL-C Ratio: Base Study | Baseline and Week 8 of Base Study
Change from Baseline in C-reactive Protein (CRP): Base Study | Baseline and Week 8 of Base Study
Percentage Change from Baseline in LDL-C: Extension | Baseline (Week 6) and Week 18 of Extension

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Masana L, Mata P, Gagne C, Sirah W, Cho M, Johnson-Levonas AO, Meehan A, Troxell JK, Gumbiner B; Ezetimibe Study Group. Long-term safety and, tolerability profiles and lipid-modifying efficacy of ezetimibe coadministered with ongoing simvastatin treatment: a multicenter, randomized, double-blind, placebo-controlled, 48-week extension study. Clin Ther. 2005 Feb;27(2):174-84. doi: 10.1016/j.clinthera.2005.02.011. PMID 15811480
- [Result] Gagne C, Bays HE, Weiss SR, Mata P, Quinto K, Melino M, Cho M, Musliner TA, Gumbiner B; Ezetimibe Study Group. Efficacy and safety of ezetimibe added to ongoing statin therapy for treatment of patients with primary hypercholesterolemia. Am J Cardiol. 2002 Nov 15;90(10):1084-91. doi: 10.1016/s0002-9149(02)02774-1. PMID 12423708